CLINICAL TRIAL: NCT06215521
Title: A Phase I, Single-Dose, Randomized, Partially Double-Blind, Placebo- and Positive-Controlled, 3-Way Crossover Study to Evaluate the Effect of LOXO-305 on QTc Interval in Healthy Subjects
Brief Title: A Study to Evaluate the Effect of Pirtobrutinib (LOXO-305) on QTc Interval in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Collaborators: Loxo Oncology, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: LOXO-BTK-20011; J2N-OX-JZNI (Other: Eli Lilly and Company)
Record Dates: First submitted 2023-12-15; First posted 2024-01-22 (Actual); Results first posted 2025-02-24 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2025-01

CONDITIONS: Healthy
MeSH Terms: interventions — pirtobrutinib; Moxifloxacin

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: This is a partially double-blind study (for LOXO-305 only, not moxifloxacin).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Pirtobrutinib (Experimental): Pirtobrutinib a single oral dose on Day 1, 12 and 23 following a fast of at least 8 hours prior to and 6 hours after dosing.
  Interventions: Drug: Pirtobrutinib
- Placebo (Placebo Comparator): Placebo (matched to Pirtobrutinib) a single oral dose on Day 1, 12 and 23 following a fast of at least 8 hours prior to and 6 hours after dosing.
  Interventions: Drug: Placebo
- Moxifloxacin (Active Comparator): Moxifloxacin a single oral dose on Day 1, 12 and 23 following a fast of at least 8 hours prior to and 6 hours after dosing.
  Interventions: Drug: Moxifloxacin

INTERVENTIONS:
Drug: Pirtobrutinib — Administered orally
  Other Names: LOXO-305; LY3527727
  Arms: Pirtobrutinib
Drug: Placebo — Administered orally
  Arms: Placebo
Drug: Moxifloxacin — Administered orally
  Arms: Moxifloxacin

SUMMARY:
The main purpose of this study is to assess the effect of Pirtobrutinib (LOXO-305) on the heart rate-corrected QT (QTc) interval and to conduct blood tests to measure how much pirtobrutinib (LOXO-305) is in the bloodstream and how the body handles and eliminates pirtobrutinib. The study will also evaluate the safety and tolerability of pirtobrutinib. The study will last up to 71 days, including screening.

ELIGIBILITY:
Inclusion Criteria:

* Must have Body mass index (BMI) within the range of 18.0 to 32.0 kilograms per square meter (kg/m²), inclusive at Screening
* Male and female participants in good health, determined by no clinically significant findings from medical history, 12-lead Electrocardiogram (ECG), vital sign measurements, or clinical laboratory evaluations as assessed by the investigator
* Female participants of non-childbearing potential and male participants who follow standard contraceptive methods
* Must have comply with all study procedures, including the 15-night stay at the Clinical Research Unit (CRU) and follow-up phone call

Exclusion Criteria:

* History or presence of any diseases or conditions of clinical significance by the Investigator (or designee) and/or Sponsor
* Positive serologic test for hepatitis B surface antigen (HBsAg), hepatitis B virus immunoglobulin M (HBV IgM) core antibody, hepatitis C virus (HCV) antibody, or human immunodeficiency virus (HIV) antibody at Screening.
* Positive polymerase chain reaction (PCR) test for COVID-19 at Screening
* Known ongoing alcohol and/or drug abuse within 2 years prior to Screening
* History of significant hypersensitivity, intolerance, or allergy to any drug compound, food, or other substance, unless approved by the Investigator (or designee)
* Have previously received pirtobrutinib (LOXO-305) in any other study investigating pirtobrutinib (LOXO-305), within 30 days prior to Day 1

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 31 (Actual)
Dates: Start 2020-12-15 (Actual); Primary Completion 2021-03-31 (Actual); Study Completion 2021-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Renee Ward, MD, PhD, Study Director — Loxo Oncology, Inc.
Locations (2):
- United States (2):
  - Covance Clinical Research Unit 1341 Mockingbird Lane, Dallas, Texas
  - Covance Clinical Research Unit 3402 Kinsman Blvd, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 31 participants were enrolled in this study. Participants were randomly assigned to 1 of 6 treatment sequences (ABC, BCA, CAB, ACB, CBA and BAC) where Treatment A was single oral dose of 900 milligrams (mg) pirtobrutinib, Treatment B was single oral dose of 900 mg pirtobrutinib matched placebo and Treatment C was single oral dose of 400 mg moxifloxacin.
Groups:
- Treatment Sequence 1: ABC: Participants received a single oral dose of 900 mg pirtobrutinib (Treatment A) on Day 1, followed by a single oral dose of 900 mg pirtobrutinib matched placebo (Treatment B) on Day 12 and a single oral dose of 400 mg moxifloxacin (Treatment C) on Day 23, under fasted conditions.
- Treatment Sequence 2: BCA: Participants received a single oral dose of 900 mg pirtobrutinib matched placebo (Treatment B) on Day 1, followed by a single oral dose of 400 mg moxifloxacin (Treatment C) on Day 12 and a single oral dose of 900 mg pirtobrutinib (Treatment A) on Day 23, under fasted conditions.
- Treatment Sequence 3: CAB: Participants received a single oral dose of 400 mg moxifloxacin (Treatment C) on Day 1, followed by a single oral dose of 900 mg pirtobrutinib (Treatment A) on Day 12 and a single oral dose of 900 mg pirtobrutinib matched placebo (Treatment B) on Day 23, under fasted conditions.
- Treatment Sequence 4: ACB: Participants received a single oral dose of 900 mg pirtobrutinib (Treatment A) on Day 1, followed by a single oral dose of 400 mg moxifloxacin (Treatment C) on Day 12 and a single oral dose of 900 mg pirtobrutinib matched placebo (Treatment B) on Day 23, under fasted conditions.
- Treatment Sequence 5: CBA: Participants received a single oral dose of 400 mg moxifloxacin (Treatment C) on Day 1, followed by a single oral dose of 900 mg pirtobrutinib matched placebo (Treatment B) on Day 12 and a single oral dose of 900 mg pirtobrutinib (Treatment A) on Day 23, under fasted conditions.
- Treatment Sequence 6: BAC: Participants received a single oral dose of 900 mg pirtobrutinib matched placebo (Treatment B) on Day 1, followed by a single oral dose of 900 mg pirtobrutinib (Treatment A) on Day 12 and a single oral dose of 400 mg moxifloxacin (Treatment C) on Day 23, under fasted conditions.
Period: Treatment Period 1 (Day 1)
Arm/Group | Treatment Sequence 1: ABC | Treatment Sequence 2: BCA | Treatment Sequence 3: CAB | Treatment Sequence 4: ACB | Treatment Sequence 5: CBA | Treatment Sequence 6: BAC
Started | 5 | 6 | 5 | 5 | 5 | 5
Received 1 Dose of Treatment A | 5 | 5 | 5 | 5 | 5 | 5
Received 1 Dose of Treatment B | 5 | 6 | 5 | 5 | 5 | 5
Received 1 Dose of Treatment C | 5 | 5 | 5 | 5 | 5 | 5
Completed | 5 | 5 | 5 | 5 | 5 | 5
Not Completed | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 1 | 0 | 0 | 0 | 0
Period: Treatment Period 2 (Day 12)
Arm/Group | Treatment Sequence 1: ABC | Treatment Sequence 2: BCA | Treatment Sequence 3: CAB | Treatment Sequence 4: ACB | Treatment Sequence 5: CBA | Treatment Sequence 6: BAC
Started | 5 | 5 | 5 | 5 | 5 | 5
Completed | 5 | 5 | 5 | 5 | 5 | 5
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Treatment Period 3 (Day 23)
Arm/Group | Treatment Sequence 1: ABC | Treatment Sequence 2: BCA | Treatment Sequence 3: CAB | Treatment Sequence 4: ACB | Treatment Sequence 5: CBA | Treatment Sequence 6: BAC
Started | 5 | 5 | 5 | 5 | 5 | 5
Completed | 5 | 5 | 5 | 5 | 5 | 5
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All participants who received 1 dose of study drug.
Groups:
- Treatment Sequence: ABC: Participants received a single oral dose of 900 mg pirtobrutinib (Treatment A) on Day 1, followed by a single oral dose of 900 mg pirtobrutinib matched placebo (Treatment B) on Day 12 and a single oral dose of 400 mg moxifloxacin (Treatment C) on Day 23, under fasted conditions
- Treatment Sequence: BCA: Participants received a single oral dose of 900 mg pirtobrutinib matched placebo (Treatment B) on Day 1, followed by a single oral dose of 400 mg moxifloxacin (Treatment C) on Day 12 and a single oral dose of 900 mg pirtobrutinib (Treatment A) on Day 23, under fasted conditions.
- Treatment Sequence: CAB: Participants received a single oral dose of 400 mg moxifloxacin (Treatment C) on Day 1, followed by a single oral dose of 900 mg pirtobrutinib (Treatment A) on Day 12 and a single oral dose of 900 mg pirtobrutinib matched placebo (Treatment B) on Day 23, under fasted conditions.
- Treatment Sequence: ACB: Participants received a single oral dose of 900 mg pirtobrutinib (Treatment A) on Day 1, followed by a single oral dose of 400 mg moxifloxacin (Treatment C) on Day 12 and a single oral dose of 900 mg pirtobrutinib matched placebo (Treatment B) on Day 23, under fasted conditions.
- Treatment Sequence: CBA: Participants received a single oral dose of 400 mg moxifloxacin (Treatment C) on Day 1, followed by a single oral dose of 900 mg pirtobrutinib matched placebo (Treatment B) on Day 12 and a single oral dose of 900 mg pirtobrutinib (Treatment A) on Day 23, under fasted conditions.
- Treatment Sequence: BAC: Participants received a single oral dose of 900 mg pirtobrutinib matched placebo (Treatment B) on Day 1, followed by a single oral dose of 900 mg pirtobrutinib (Treatment A) on Day 12 and a single oral dose of 400 mg moxifloxacin (Treatment C) on Day 23, under fasted conditions.
- Total: Total of all reporting groups
Arm/Group | Treatment Sequence: ABC | Treatment Sequence: BCA | Treatment Sequence: CAB | Treatment Sequence: ACB | Treatment Sequence: CBA | Treatment Sequence: BAC | Total
Number analyzed (Participants) | 5 | 6 | 5 | 5 | 5 | 5 | 31
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.0 (9.87) | 39.0 (8.81) | 37.8 (7.95) | 35.6 (7.86) | 34.4 (6.77) | 38.2 (10.01) | 36.7 (8.08)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 2 | 0 | 0 | 2 | 7
  Male | 4 | 4 | 3 | 5 | 5 | 3 | 24
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1 | 2 | 1 | 3 | 8
  Not Hispanic or Latino | 4 | 6 | 4 | 3 | 4 | 2 | 23
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 1 | 0 | 0 | 1
  Asian | 1 | 0 | 0 | 0 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 1 | 0 | 1
  Black or African American | 4 | 4 | 2 | 1 | 1 | 2 | 14
  White | 0 | 2 | 3 | 3 | 3 | 3 | 14
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 5 | 6 | 5 | 5 | 5 | 5 | 31

OUTCOME MEASURES:

1. Primary Outcome: Placebo-corrected Change From Baseline in QT Interval Corrected Using Fridericia's Correction (QTcF) (ΔΔQTcF)
Description: The cardiodynamic assessment was performed through 12-lead electrocardiogram (ECG) extracted from continuous recordings at pre-specified time points. Participants rested in supine position for at least 10 minutes prior to and 5 minutes after each time point for ECG extractions. The QT interval is the time from electrocardiogram Q wave to the end of the T wave corresponding to electrical systole. QT interval was corrected for heart rate using QTcF. Placebo-corrected change from baseline in QTcF (ΔΔQTcF) was calculated based on model-predicted effect.
Time Frame: Baseline (Predose), 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8.5, 12 and 24 hours post-dose
Population: Pharmacokinetic/Corrected QT interval (PK/QTc) population included all participants who were in both the PK and QT/QTc populations with at least 1 pair of post-dose PK and ΔQTc data from the same time point in at least 1 period as well as participants in the QT/QTc population who received placebo. As per planned analysis, data was planned to be reported only for Treatment A (900 mg pirtobrutinib) concentration for this outcome measure.
Measure: Least Squares Mean (90% Confidence Interval); unit: milliseconds (msec)
Groups:
- Treatment A: 900 mg Pirtobrutinib: Participants who received a single oral dose of 900 mg Pirtobrutinib capsules.
Arm/Group | Treatment A: 900 mg Pirtobrutinib
Number analyzed (Participants) | 30
milliseconds (msec) | 0.73 [-1.17 to 2.64]

2. Secondary Outcome: Change From Baseline in (Δ) QTcF
Description: The cardiodynamic assessment was performed through 12-lead ECG extracted from continuous recordings at pre-specified time points. Participants rested in supine position for at least 10 minutes prior to and 5 minutes after each time point for ECG extractions. The QT interval is the time from electrocardiogram Q wave to the end of the T wave corresponding to electrical systole. QT interval was corrected for heart rate using QTcF. Change from baseline in (Δ) QTcF was calculated using linear mixed-effects model analysis.
Time Frame: Baseline (predose), 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8.5, 12 and 24 hours post-dose
Population: QT/QTc population included all participants who received 1 dose of study drug with measurements at baseline as well as on treatment with at least 1 post-dose time point with a valid ΔQTc value. Here, 'Number Analyzed' signifies participants who were evaluable at specific timepoints.
Measure: Least Squares Mean (90% Confidence Interval); unit: msec
Groups:
- Treatment A: 900 mg Pirtobrutinib: Participants who received a single oral dose of 900 mg pirtobrutinib capsule.
- Treatment B: 900 mg Pirtobrutinib Matched Placebo: Participants who received a single oral dose of 900 mg pirtobrutinib matched placebo capsules.
- Treatment C: 400 mg Moxifloxacin: Participants who received a single oral dose of 400 mg moxifloxacin tablets.
Arm/Group | Treatment A: 900 mg Pirtobrutinib | Treatment B: 900 mg Pirtobrutinib Matched Placebo | Treatment C: 400 mg Moxifloxacin
Number analyzed (Participants) | 30 | 30 | 29
msec
  Change at 0.25 hour post-dose | -0.4 [-1.41 to 0.68] | 0.0 [-1.01 to 1.08] | -0.1 [-1.15 to 0.97]
  Change at 0.5 hour post-dose | -4.5 [-5.94 to -3.06] | -2.8 [-4.21 to -1.33] | 4.2 [2.72 to 5.66]
  Change at 0.75 hour post-dose | -3.8 [-5.37 to -2.29] | -2.0 [-3.50 to -0.42] | 7.6 [6.03 to 9.17]
  Change at 1 hour post-dose: number analyzed (Participants) | 27 | 28 | 28
  Change at 1 hour post-dose | -2.8 [-4.25 to -1.33] | -1.2 [-2.65 to 0.24] | 8.3 [6.88 to 9.80]
  Change at 1.5 hours post-dose | -0.6 [-2.26 to 0.98] | -1.0 [-2.63 to 0.61] | 9.8 [8.15 to 11.45]
  Change at 2 hours post-dose | -2.2 [-3.89 to -0.49] | -1.1 [-2.80 to 0.60] | 9.4 [7.64 to 11.10]
  Change at 2.5 hours post-dose | -0.2 [-1.89 to 1.46] | 0.2 [-1.45 to 1.90] | 10.1 [8.39 to 11.82]
  Change at 3 hours post-dose: number analyzed (Participants) | 30 | 30 | 28
  Change at 3 hours post-dose | 0.3 [-1.45 to 2.13] | 0.5 [-1.26 to 2.32] | 9.9 [8.11 to 11.75]
  Change at 4 hours post-dose | 2.2 [0.18 to 4.19] | 0.3 [-1.70 to 2.32] | 9.8 [7.78 to 11.86]
  Change at 6 hours post-dose | 3.5 [1.48 to 5.42] | 0.9 [-1.08 to 2.86] | 9.3 [7.26 to 11.26]
  Change at 8.5 hours post-dose | -5.1 [-7.07 to -3.09] | -5.2 [-7.15 to -3.17] | 2.8 [0.80 to 4.85]
  Change at 12 hours post-dose: number analyzed (Participants) | 30 | 30 | 28
  Change at 12 hours post-dose | 1.2 [-1.41 to 3.75] | 0.6 [-1.99 to 3.17] | 6.8 [4.12 to 9.44]
  Change at 24 hours post-dose: number analyzed (Participants) | 30 | 28 | 28
  Change at 24 hours post-dose | 0.0 [-1.71 to 1.69] | 0.6 [-1.11 to 2.41] | 5.0 [3.22 to 6.74]

3. Secondary Outcome: Change From Baseline in Heart Rate (ΔHR)
Description: Heart rate is the number of times the ventricles of the heart contract and relax per minute. Change from baseline in heart rate (ΔHR) was calculated using linear mixed-effects model analysis.
Time Frame: Baseline (predose), 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8.5, 12 and 24 hours post-dose
Population: QT/QTc population included all participants who received 1 dose of study drug with measurements at baseline as well as on treatment with at least 1 post-dose time point with a valid ΔQTc value. Here, 'Number Analyzed' signifies participants who were evaluable at specific timepoints. As per planned analysis, data was planned to be reported only for Treatment A and B for this outcome measure.
Measure: Least Squares Mean (90% Confidence Interval); unit: beats per minute (beats/min)
Arm/Group | Treatment A: 900 mg Pirtobrutinib | Treatment B: 900 mg Pirtobrutinib Matched Placebo
Number analyzed (Participants) | 30 | 30
beats per minute (beats/min)
  Change at 0.25 hour post-dose | 0.1 [-0.94 to 1.07] | -0.9 [-1.81 to 0.09]
  Change at 0.5 hour post-dose | -0.5 [-1.66 to 0.61] | -1.2 [-2.24 to -0.07]
  Change at 0.75 hour post-dose | 0.0 [-1.28 to 1.23] | -0.4 [-1.66 to 0.76]
  Change at 1 hour post-dose: number analyzed (Participants) | 27 | 28
  Change at 1 hour post-dose | 1.0 [-0.23 to 2.32] | -0.1 [-1.34 to 1.09]
  Change at 1.5 hours post-dose | 0.9 [-0.28 to 2.06] | -1.7 [-2.82 to -0.58]
  Change at 2 hours post-dose | 0.5 [-0.73 to 1.76] | -0.8 [-1.98 to 0.42]
  Change at 2.5 hours post-dose | 2.2 [0.87 to 3.54] | -0.1 [-1.37 to 1.22]
  Change at 3 hours post-dose | 1.3 [-0.01 to 2.52] | 0.4 [-0.84 to 1.60]
  Change at 4 hours post-dose | 1.4 [0.12 to 2.67] | 0.4 [-0.85 to 1.61]
  Change at 6 hours post-dose | 2.0 [0.65 to 3.43] | 0.5 [-0.88 to 1.82]
  Change at 8.5 hours post-dose | 4.0 [2.42 to 5.59] | 3.4 [1.89 to 5.00]
  Change at 12 hours post-dose | 2.0 [0.22 to 3.74] | 0.4 [-1.36 to 2.09]
  Change at 24 hours post-dose: number analyzed (Participants) | 30 | 28
  Change at 24 hours post-dose | 1.2 [0.00 to 2.48] | 0.8 [-0.41 to 2.04]

4. Secondary Outcome: Change From Baseline in Pulse Rate (ΔPR)
Description: Pulse rate is number of times heart beats per minute. Pulse rate measurements were performed using the same arm for each reading and measurements were taken after the participant had been resting in the supine position for at least 5 minutes. Change from baseline in pulse rate (ΔPR) was calculated using linear mixed-effects model analysis.
Time Frame: Baseline (predose), 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8.5, 12 and 24 hours post-dose
Population: QT/QTc population included all participants who received 1 dose of study drug with measurements at baseline as well as on treatment with at least 1 post-dose time point with a valid ΔQTc value. Here, 'Number Analyzed' signifies participants evaluable for specific timepoints. As per planned analysis, data was planned to be reported only for Treatment A and B for this outcome measure.
Measure: Least Squares Mean (90% Confidence Interval); unit: beats per minute (beats/min)
Arm/Group | Treatment A: 900 mg Pirtobrutinib | Treatment B: 900 mg Pirtobrutinib Matched Placebo
Number analyzed (Participants) | 30 | 30
beats per minute (beats/min)
  Change at 0.25 hour post-dose | -2.6 [-4.46 to -0.83] | -0.8 [-2.60 to 1.02]
  Change at 0.5 hour post-dose | 0.3 [-1.61 to 2.15] | 1.5 [-0.42 to 3.34]
  Change at 0.75 hour post-dose | 0.3 [-1.41 to 1.98] | 1.0 [-0.72 to 2.67]
  Change at 1 hour post-dose: number analyzed (Participants) | 27 | 28
  Change at 1 hour post-dose | -0.1 [-2.24 to 2.11] | 0.7 [-1.48 to 2.83]
  Change at 1.5 hours post-dose | -0.9 [-2.69 to 0.81] | -1.2 [-2.96 to 0.54]
  Change at 2 hours post-dose | -0.5 [-1.97 to 0.99] | -0.5 [-1.94 to 1.01]
  Change at 2.5 hours post-dose | -3.9 [-5.82 to -2.02] | -0.8 [-2.73 to 1.06]
  Change at 3 hours post-dose | -0.9 [-2.87 to 1.13] | -1.3 [-3.30 to 0.70]
  Change at 4 hours post-dose | -1.6 [-3.23 to 0.05] | -2.3 [-3.91 to -0.64]
  Change at 6 hours post-dose | -4.4 [-6.12 to -2.73] | -2.7 [-4.34 to -0.96]
  Change at 8.5 hours post-dose | -6.2 [-8.30 to -4.06] | -5.1 [-7.24 to -3.00]
  Change at 12 hours post-dose | -4.9 [-7.82 to -1.88] | -2.8 [-5.77 to 0.17]
  Change at 24 hours post-dose: number analyzed (Participants) | 30 | 28
  Change at 24 hours post-dose | -4.2 [-6.59 to -1.75] | -0.6 [-3.11 to 1.90]

5. Secondary Outcome: Change From Baseline in QRS Intervals (Δ QRS)
Description: QRS interval in an ECG measured the total time of ventricular depolarization. It begins with Q or R wave and ends at the end of the S wave. Change from baseline in QRS intervals (Δ QRS) was calculated using linear mixed-effects model analysis.
Time Frame: Baseline (predose), 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8.5, 12 and 24 hours post-dose
Population: as for outcome 4
Measure: Least Squares Mean (90% Confidence Interval); unit: msec
Groups:
- Treatment B: Pirtobrutinib Matched Placebo: Participants who received a single oral dose of pirtobrutinib matched placebo capsules.
Arm/Group | Treatment A: 900 mg Pirtobrutinib | Treatment B: Pirtobrutinib Matched Placebo
Number analyzed (Participants) | 30 | 30
msec
  Change at 0.25 hour post-dose | 0.0 [-0.24 to 0.24] | 0.0 [-0.26 to 0.22]
  Change at 0.5 hour post-dose | 0.2 [-0.03 to 0.45] | -0.1 [-0.37 to 0.11]
  Change at 0.75 hour post-dose | 0.2 [-0.01 to 0.42] | 0.0 [-0.18 to 0.25]
  Change at 1 hour post-dose: number analyzed (Participants) | 27 | 28
  Change at 1 hour post-dose | 0.2 [-0.18 to 0.49] | -0.1 [-0.43 to 0.22]
  Change at 1.5 hours post-dose | -0.1 [-0.34 to 0.17] | -0.1 [-0.35 to 0.15]
  Change at 2 hours post-dose | 0.0 [-0.29 to 0.20] | -0.1 [-0.33 to 0.16]
  Change at 2.5 hours post-dose | -0.1 [-0.39 to 0.18] | -0.1 [-0.41 to 0.15]
  Change at 3 hours post-dose | 0.2 [-0.06 to 0.50] | -0.1 [-0.38 to 0.18]
  Change at 4 hours post-dose | 0.2 [-0.13 to 0.44] | 0.1 [-0.19 to 0.37]
  Change at 6 hours post-dose | 0.7 [0.30 to 1.01] | 0.2 [-0.19 to 0.52]
  Change at 8.5 hours post-dose | -0.6 [-1.17 to -0.12] | 0.1 [-0.42 to 0.63]
  Change at 12 hours post-dose | 0.4 [-0.11 to 0.83] | 0.3 [-0.16 to 0.78]
  Change at 24 hours post-dose: number analyzed (Participants) | 30 | 28
  Change at 24 hours post-dose | 0.2 [-0.81 to 1.23] | -1.0 [-2.03 to 0.10]

6. Secondary Outcome: Change From Baseline in Individualized Heart Rate-Corrected QT Interval (ΔQTcS), If a Substantial Heart Rate Effect Was Observed
Description: The cardiodynamic assessment was performed through 12-lead ECG extracted from continuous recordings at pre-specified time points. Participants rested in supine position for at least 10 minutes prior to and 5 minutes after each time point for ECG extractions. The QT interval is the time from electrocardiogram Q wave to the end of the T wave corresponding to electrical systole. QT interval was corrected for heart rate using QTcS.
Time Frame: Baseline (predose), 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8.5, 12 and 24 hours post-dose
Population: QT/QTc population included all participants who received 1 dose of study drug with measurements at baseline as well as on treatment with at least 1 post-dose time point with a valid ΔQTc value. As per planned analysis, data was planned to be reported only for Treatment A and B for this outcome measure.
Measure: Least Squares Mean (90% Confidence Interval); unit: msec
Groups:
- Treatment B: Pirtobrutinib Matched Placebo: Participants who received a single oral dose of 900 mg pirtobrutinib matched placebo capsules.
Arm/Group | Treatment A: 900 mg Pirtobrutinib | Treatment B: Pirtobrutinib Matched Placebo
Number analyzed (Participants) | 30 | 30
msec | NA [NA to NA] — Pirtobrutinib did not cause a substantial HR effect, the Fridericia's formula was chosen as the HR correction method for the QT analysis and hence the other QT correction methods (QTcS with hysteresis adjustment) could not be calculated. | NA [NA to NA] — Pirtobrutinib Matched Placebo did not cause a substantial HR effect, the Fridericia's formula was chosen as the HR correction method for the QT analysis and hence the other QT correction methods (QTcS with hysteresis adjustment) could not be calculated.

7. Secondary Outcome: Change From Baseline in Optimized Heart Rate-Corrected QT Interval (ΔQTcI), If a Substantial Heart Rate Effect Was Observed
Description: The cardiodynamic assessment was performed through 12-lead ECG extracted from continuous recordings at pre-specified time points. Participants rested in supine position for at least 10 minutes prior to and 5 minutes after each time point for ECG extractions. The QT interval is the time from electrocardiogram Q wave to the end of the T wave corresponding to electrical systole. QT interval was corrected for heart rate using QTcI.
Time Frame: Baseline (predose), 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8.5, 12 and 24 hours post-dose
Population: as for outcome 6
Measure: Least Squares Mean (90% Confidence Interval); unit: msec
Arm/Group | Treatment A: 900 mg Pirtobrutinib | Treatment B: Pirtobrutinib Matched Placebo
Number analyzed (Participants) | 30 | 30
msec | NA [NA to NA] — Pirtobrutinib did not cause a substantial HR effect, the Fridericia's formula was chosen as the HR correction method for the QT analysis and hence the other QT correction methods (QTcI with hysteresis adjustment) could not be calculated. | NA [NA to NA] — Pirtobrutinib matched placebo did not cause a substantial HR effect, the Fridericia's formula was chosen as the HR correction method for the QT analysis and hence the other QT correction methods (QTcI with hysteresis adjustment) could not be calculated.

8. Secondary Outcome: Placebo-corrected Change From Baseline in Heart Rate (ΔΔHR)
Description: Heart rate is the number of times the ventricles of the heart contract and relax per minute. Placebo-corrected change from baseline in heart rate (ΔΔHR) was calculated using linear mixed-effects model analysis.
Time Frame: Baseline (predose), 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8.5, 12 and 24 hours post-dose
Population: QT/QTc population included all participants who received 1 dose of study drug with measurements at baseline as well as on treatment with at least 1 post-dose time point with a valid ΔQTc value. As per planned analysis, data was planned to be reported only for Treatment A and C for this outcome measure.
Measure: Least Squares Mean (90% Confidence Interval); unit: beats/min
Arm/Group | Treatment A: 900 mg Pirtobrutinib | Treatment C: 400 mg Moxifloxacin
Number analyzed (Participants) | 30 | 29
beats/min
  Change at 0.25 hours post-dose | 0.9 [-0.11 to 1.96] | 0.1 [-0.92 to 1.15]
  Change at 0.5 hours post-dose | 0.6 [-0.65 to 1.90] | 3.0 [1.71 to 4.27]
  Change at 0.75 hours post-dose | 0.4 [-1.06 to 1.91] | 3.8 [2.35 to 5.34]
  Change at 1 hour post-dose | 1.2 [-0.33 to 2.68] | 4.2 [2.71 to 5.71]
  Change at 1.5 hours post-dose | 2.6 [1.26 to 3.92] | 2.8 [1.43 to 4.10]
  Change at 2 hours post-dose | 1.3 [-0.18 to 2.77] | 2.5 [1.02 to 3.99]
  Change at 2.5 hours post-dose | 2.3 [0.66 to 3.90] | 2.9 [1.25 to 4.53]
  Change at 3 hours post-dose | 0.9 [-0.63 to 2.38] | 1.1 [-0.38 to 2.65]
  Change at 4 hours post-dose | 1.0 [-0.51 to 2.53] | 1.9 [0.34 to 3.40]
  Change at 6 hours post-dose | 1.6 [-0.14 to 3.28] | 2.6 [0.86 to 4.32]
  Change at 8.5 hours post-dose | 0.6 [-1.47 to 2.58] | 1.5 [-0.54 to 3.54]
  Change at 12 hours post-dose | 1.6 [-0.68 to 3.91] | 4.5 [2.16 to 6.82]
  Change at 24 hours post-dose | 0.4 [-1.06 to 1.91] | 1.0 [-0.47 to 2.54]

9. Secondary Outcome: Placebo-corrected Change From Baseline in Pulse Rate (ΔΔ PR)
Description: Pulse rate is number of times heart beats per minute. Pulse rate measurements were performed using the same arm for each reading and measurements were taken after the participant had been resting in the supine position for at least 5 minutes. Placebo-corrected change from baseline in pulse rate (ΔPR) was calculated using linear mixed-effects model analysis.
Time Frame: Baseline (predose), 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8.5, 12 and 24 hours post-dose
Population: as for outcome 8
Measure: Least Squares Mean (90% Confidence Interval); unit: beats/min
Arm/Group | Treatment A: 900 mg Pirtobrutinib | Treatment C: 400 mg Moxifloxacin
Number analyzed (Participants) | 30 | 29
beats/min
  Change at 0.25 hours post-dose | -1.9 [-4.28 to 0.56] | -1.2 [-3.65 to 1.24]
  Change at 0.5 hours post-dose | -1.2 [-3.72 to 1.33] | -2.1 [-4.68 to 0.42]
  Change at 0.75 hours post-dose | -0.7 [-2.93 to 1.55] | -2.5 [-4.80 to -0.27]
  Change at 1 hours post-dose | -0.7 [-3.69 to 2.20] | -3.8 [-6.78 to -0.88]
  Change at 1.5 hours post-dose | 0.3 [-2.05 to 2.60] | -3.4 [-5.78 to -1.09]
  Change at 2 hours post-dose | 0.0 [-1.94 to 1.89] | -3.6 [-5.54 to -1.68]
  Change at 2.5 hours post-dose | -3.1 [-5.64 to -0.54] | -4.6 [-7.23 to -2.05]
  Change at 3 hours post-dose | 0.4 [-2.27 to 3.13] | -4.0 [-6.70 to -1.26]
  Change at 4 hours post-dose | 0.7 [-1.47 to 2.85] | -4.2 [-6.33 to -1.98]
  Change at 6 hours post-dose | -1.8 [-4.01 to 0.47] | -4.3 [-6.53 to -2.02]
  Change at 8.5 hours post-dose | -1.1 [-3.94 to 1.82] | -2.1 [-5.00 to 0.80]
  Change at 12 hours post-dose | -2.1 [-6.17 to 2.06] | -3.5 [-7.63 to 0.71]
  Change at 24 hours post-dose | -3.6 [-6.95 to -0.18] | -0.8 [-4.19 to 2.69]

10. Secondary Outcome: Placebo-Corrected Change From Baseline in QRS (ΔΔQRS)
Description: QRS interval in an ECG measured the total time of ventricular depolarization. It begins with Q or R wave and ends at the end of the S wave. Placebo-corrected change from baseline in QRS intervals (ΔΔQRS) was calculated using linear mixed-effects model analysis.
Time Frame: Baseline (predose), 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8.5, 12 and 24 hours post-dose
Population: as for outcome 8
Measure: Least Squares Mean (90% Confidence Interval); unit: msec
Arm/Group | Treatment A: 900 mg Pirtobrutinib | Treatment C: 400 mg Moxifloxacin
Number analyzed (Participants) | 30 | 29
msec
  Change at 0.25 hours post-dose | 0.0 [-0.32 to 0.36] | -0.3 [-0.63 to 0.06]
  Change at 0.5 hours post-dose | 0.3 [0.00 to 0.68] | 0.1 [-0.26 to 0.43]
  Change at 0.75 hours post-dose | 0.2 [-0.13 to 0.47] | 0.3 [0.03 to 0.63]
  Change at 1 hours post-dose | 0.3 [-0.21 to 0.73] | 0.1 [-0.34 to 0.59]
  Change at 1.5 hours post-dose | 0.0 [-0.34 to 0.37] | 0.1 [-0.22 to 0.49]
  Change at 2 hours post-dose | 0.0 [-0.30 to 0.39] | 0.1 [-0.20 to 0.50]
  Change at 2.5 hours post-dose | 0.0 [-0.37 to 0.43] | 0.1 [-0.33 to 0.48]
  Change at 3 hours post-dose | 0.3 [-0.07 to 0.72] | -0.1 [-0.50 to 0.29]
  Change at 4 hours post-dose | 0.1 [-0.33 to 0.46] | -0.3 [-0.67 to 0.13]
  Change at 6 hours post-dose | 0.5 [-0.01 to 0.99] | -0.1 [-0.58 to 0.43]
  Change at 8.5 hours post-dose | -0.8 [-1.50 to -0.01] | -0.4 [-1.12 to 0.38]
  Change at 12 hours post-dose | 0.1 [-0.62 to 0.72] | 0.0 [-0.65 to 0.70]
  Change at 24 hours post-dose | 1.2 [-0.30 to 2.65] | 0.2 [-1.25 to 1.74]

11. Secondary Outcome: Placebo-corrected Change From Baseline in ΔQTcF (ΔΔQTcF), If a Substantial Heart Rate Effect Was Observed
Description: The cardiodynamic assessment was performed through 12-lead ECG extracted from continuous recordings at pre-specified time points. Participants rested in supine position for at least 10 minutes prior to and 5 minutes after each time point for ECG extractions. The QT interval is the time from electrocardiogram Q wave to the end of the T wave corresponding to electrical systole. QT interval was corrected for heart rate using QTcF.
Time Frame: Baseline (predose), 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8.5, 12 and 24 hours post-dose
Population: PK/QTc population included all participants who were in both the PK and QT/QTc populations with at least 1 pair of post-dose PK and ΔQTc data from the same time point in at least 1 period as well as participants in the QT/QTc population who received placebo. As per planned analysis, data was planned to be reported only for Treatment A and B for this outcome measure.
Measure: Least Squares Mean (90% Confidence Interval); unit: msec
Arm/Group | Treatment A: 900 mg Pirtobrutinib | Treatment B: 900 mg Pirtobrutinib Matched Placebo
Number analyzed (Participants) | 30 | 30
msec | NA [NA to NA] — Pirtobrutinib did not cause a substantial HR effect, hence data could not be calculated. | NA [NA to NA] — Pirtobrutinib matched placebo did not cause a substantial HR effect, hence data could not be calculated.

12. Secondary Outcome: Placebo-corrected Change From Baseline in Individualized Heart Rate-Corrected QT Interval (ΔΔQTcS), If a Substantial Heart Rate Effect Was Observed
Description: as for outcome 6
Time Frame: Baseline (predose), 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8.5, 12 and 24 hours post-dose
Population: QT/QTc population included all participants w.ho received 1 dose of study drug with measurements at baseline as well as on treatment with at least 1 post-dose time point with a valid ΔQTc value. As per planned analysis, data was planned to be reported only for Treatment A and B for this outcome measure
Measure: Least Squares Mean (90% Confidence Interval); unit: msec
Arm/Group | Treatment A: 900 mg Pirtobrutinib | Treatment B: 900 mg Pirtobrutinib Matched Placebo
Number analyzed (Participants) | 30 | 30
msec | NA [NA to NA] — Pirtobrutinib did not cause a substantial HR effect, the Fridericia's formula was chosen as the HR correction method for the QT analysis and hence the other QT correction methods (QTcS with hysteresis adjustment) could not be calculated. | NA [NA to NA] — Pirtobrutinib matched placebo did not cause a substantial HR effect, the Fridericia's formula was chosen as the HR correction method for the QT analysis and hence the other QT correction methods (QTcS with hysteresis adjustment) could not be calculated.

13. Secondary Outcome: Placebo-corrected Change From Baseline in Optimized Heart Rate-Corrected QT Interval (ΔΔQTcI), If a Substantial Heart Rate Effect Was Observed
Description: as for outcome 7
Time Frame: Baseline (predose), 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8.5, 12 and 24 hours post-dose
Population: as for outcome 6
Measure: Least Squares Mean (90% Confidence Interval); unit: msec
Arm/Group | Treatment A: 900 mg Pirtobrutinib | Treatment B: 900 mg Pirtobrutinib Matched Placebo
Number analyzed (Participants) | 30 | 30
msec | NA [NA to NA] — Pirtobrutinib did not cause a substantial HR effect, the Fridericia's formula was chosen as the HR correction method for the QT analysis and hence the other QT correction methods (QTcI with hysteresis adjustment) could not be calculated. | NA [NA to NA] — Pirtobrutinib matched placebo did not cause a substantial HR effect, the Fridericia's formula was chosen as the HR correction method for the QT analysis and hence the other QT correction methods (QTcI with hysteresis adjustment) could not be calculated.

14. Secondary Outcome: Number of Participants With Potentially Clinically Significant Electrocardiogram (ECG) Changes
Description: The cardiodynamic assessment was performed through 12-lead ECG extracted from continuous recordings at pre-specified time points. Participants rested in supine position for at least 10 minutes prior to and 5 minutes after each time point for ECG extractions. Number of participants with potentially clinically significant ECG changes were reported.
Time Frame: Baseline up to Day 33
Population: The safety population included all participants who received 1 dose of study drug. As per planned analysis, data was planned to be reported only for Treatment A and B for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment A: 900 mg Pirtobrutinib | Treatment B: 900 mg Pirtobrutinib Matched Placebo
Number analyzed (Participants) | 30 | 31
Participants | 0 | 0

15. Secondary Outcome: Number of Participants With Treatment Emergent Changes in T-wave Morphology and U-wave Presence
Description: The cardiodynamic assessment was performed through 12-lead ECG extracted from continuous recordings at pre-specified time points. Participants rested in supine position for at least 10 minutes prior to and 5 minutes after each time point for ECG extractions. Number of participants with treatment emergent changes in T-wave morphology and U-wave presence were reported.
Time Frame: Baseline up to Day 33
Population: as for outcome 14
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment A: 900 mg Pirtobrutinib | Treatment B: 900 mg Pirtobrutinib Matched Placebo
Number analyzed (Participants) | 30 | 31
Participants
  Treatment Emergent Changes in T-wave Morphology | 0 | 0
  Treatment Emergent Changes in U-wave Presence | 0 | 0

16. Secondary Outcome: Pharmacokinetic (PK): Percentage of AUC0-inf Extrapolated (AUC%Extrap) of Pirtobrutinib
Description: PK: %AUCextrap was defined as percentage extrapolation for AUC0-inf.
Time Frame: Pre-dose and 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8.5, 12, 24, 48, 72, and 96 hours post-dose
Population: PK population included participants who received 1 dose of pirtobrutinib and have at least 1 quantifiable plasma concentration of pirtobrutinib and have evaluable PK data. As per planned analysis, data was planned to be reported only for Treatment A for this outcome measure.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: percentage of AUC
Arm/Group | Treatment A: 900 mg Pirtobrutinib
Number analyzed (Participants) | 30
percentage of AUC | 5.41 (42.0)

17. Secondary Outcome: PK: Mean Residence Time (MRT) of Pirtobrutinib
Description: PK: MRT was calculated by the area under the first moment curve divided by the area under the concentration time curve.
Time Frame: Pre-dose and 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8.5, 12, 24, 48, 72, and 96 hours post-dose
Population: as for outcome 16
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | Treatment A: 900 mg Pirtobrutinib
Number analyzed (Participants) | 30
hours | 33.6 (14.6)

18. Secondary Outcome: PK: Apparent Volume of Distribution at the Terminal Phase (Vz/F) of Pirtobrutinib
Description: PK: Vz/F was defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired plasma concentration of a drug. Vz/F was calculated as (CL/F)/Lambda Z. Where, CL/F is the apparent total clearance and lambda Z is the apparent terminal elimination rate constant.
Time Frame: Pre-dose and 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8.5, 12, 24, 48, 72, and 96 hours post-dose
Population: as for outcome 16
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liter
Arm/Group | Treatment A: 900 mg Pirtobrutinib
Number analyzed (Participants) | 30
liter | 62.1 (22.5)

19. Secondary Outcome: PK: Time to Maximum Observed Plasma Concentration (Tmax) of Pirtobrutinib
Description: PK: Tmax was defined as the time to reach maximum observed plasma concentration (Cmax) for pirtobrutinib.
Time Frame: Pre-dose and 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8.5, 12, 24, 48, 72, and 96 hours post-dose
Population: as for outcome 16
Measure: Median (Full Range); unit: hours
Arm/Group | Treatment A: 900 mg Pirtobrutinib
Number analyzed (Participants) | 30
hours | 4.01 [3.00 to 24.0]

20. Secondary Outcome: PK: Apparent Plasma Terminal Elimination Half-life (t1/2) of Pirtobrutinib
Description: PK: t1/2 was defined as the terminal elimination phase half-life for pirtobrutinib.
Time Frame: Pre-dose and 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8.5, 12, 24, 48, 72, and 96 hours post-dose
Population: as for outcome 16
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | Treatment A: 900 mg Pirtobrutinib
Number analyzed (Participants) | 30
hours | 23.0 (14.5)

21. Secondary Outcome: PK: Maximum Observed Concentration (Cmax) of Pirtobrutinib
Description: PK: Cmax was defined as the maximum plasma concentration for pirtobrutinib.
Time Frame: Pre-dose and 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8.5, 12, 24, 48, 72, and 96 hours post-dose
Population: as for outcome 16
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter (ng/mL)
Arm/Group | Treatment A: 900 mg Pirtobrutinib
Number analyzed (Participants) | 30
nanogram per milliliter (ng/mL) | 14300 (23.1)

22. Secondary Outcome: PK: Area Under the Concentration-time Curve, From Time 0 to 24 Hours Post-dose (AUC0-24) of Pirtobrutinib
Description: PK: AUC(0-24) was defined as the area under the plasma concentration-time curve from 0 time to 24 hours post-dose.
Time Frame: Pre-dose and 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8.5, 12, 24 hours post-dose
Population: as for outcome 16
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour*nanogram per milliliter (h*ng/mL)
Groups:
- Treatment A: 900 mg Pirtobrutinib: Participants received a single oral dose of 900 mg pirtobrutinib capsules.
Arm/Group | Treatment A: 900 mg Pirtobrutinib
Number analyzed (Participants) | 30
hour*nanogram per milliliter (h*ng/mL) | 229000 (17.5)

23. Secondary Outcome: PK: Area Under the Concentration-time Curve, From Time 0 to the Last Measurable Concentration (AUC0-t) of Pirtobrutinib
Description: PK: AUC(0-t) was defined as the area under the plasma concentration-time curve from 0 time to last measurable point for pirtobrutinib.
Time Frame: Pre-dose and 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8.5, 12, 24, 48, 72, and 96 hours post-dose
Population: as for outcome 16
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Treatment A: 900 mg Pirtobrutinib
Number analyzed (Participants) | 30
h*ng/mL | 452000 (20.7)

24. Secondary Outcome: PK: Apparent Systemic Clearance (CL/F) of Pirtobrutinib
Description: PK: Clearance of a drug is a measure of the rate at which a drug is metabolized or eliminated by normal biological processes. CL/F was calculated as (Dose/AUC(0-inf))/F. Where AUC(0-inf) is the area under the plasma concentration-time curve from zero to infinity and F is the bioavailability of the drug.
Time Frame: Pre-dose and 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8.5, 12, 24, 48, 72, and 96 hours post-dose
Population: as for outcome 16
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liter per hour (L/h)
Arm/Group | Treatment A: 900 mg Pirtobrutinib
Number analyzed (Participants) | 30
liter per hour (L/h) | 1.88 (21.4)

25. Secondary Outcome: PK: Area Under the Concentration-time Curve From Time 0 Extrapolated to Infinity (AUC0-inf) of Pirtobrutinib
Description: PK: AUC(0-inf) was defined as the area under the plasma concentration-time curve from 0 to infinity for pirtobrutinib.
Time Frame: Pre-dose and 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8.5, 12, 24, 48, 72, and 96 hours post-dose
Population: as for outcome 16
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Treatment A: 900 mg Pirtobrutinib
Number analyzed (Participants) | 30
h*ng/mL | 480000 (21.4)

26. Secondary Outcome: PK: Apparent Terminal Elimination Rate Constant (λZ) of Pirtobrutinib
Description: PK: Terminal elimination rate constant, calculated as the negative of the slope of the log-linear regression of the natural logarithm concentration-time curve during the terminal phase.
Time Frame: Pre-dose and 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8.5, 12, 24, 48, 72, and 96 hours post-dose
Population: PK population included participants who received 1 dose of pirtobrutinib and have at least 1 quantifiable plasma concentration of pirtobrutinib and have evaluable PK data. Here, 'Overall Number of participants analyzed' signifies individual participants who were evaluable for rate constant evaluation. As per planned analysis, data was planned to be reported only for Treatment A for this outcome measure.
Measure: Number; unit: one per hour (1/h)
Arm/Group | Treatment A: 900 mg Pirtobrutinib
Number analyzed (Participants) | 30
one per hour (1/h)
  Participant 1 | 0.0320
  Participant 2 | 0.0270
  Participant 3 | 0.0356
  Participant 4 | 0.0259
  Participant 5 | 0.0270
  Participant 6 | 0.0330
  Participant 7 | 0.0310
  Participant 8 | 0.0331
  Participant 9 | 0.0353
  Participant 10 | 0.0322
  Participant 11 | 0.0271
  Participant 12 | 0.0213
  Participant 13 | 0.0337
  Participant 14 | 0.0273
  Participant 15 | 0.0229
  Participant 16 | 0.0314
  Participant 17 | 0.0364
  Participant 18 | 0.0289
  Participant 19 | 0.0309
  Participant 20 | 0.0271
  Participant 21 | 0.0269
  Participant 22 | 0.0422
  Participant 23 | 0.0346
  Participant 24 | 0.0273
  Participant 25 | 0.0288
  Participant 26 | 0.0306
  Participant 27 | 0.0364
  Participant 28 | 0.0299
  Participant 29 | 0.0304
  Participant 30 | 0.0283

ADVERSE EVENTS:
Time Frame: Baseline up to follow-up (up to Day 42)
Description: All participants who received 1 dose of study drug.
Groups:
- Treatment C: 400 mg Moxifloxacin: Participants who received a single oral dose of 400 mg Moxifloxacin tablet.
Arm/Group | Treatment A: 900 mg Pirtobrutinib | Treatment B: 900 mg Pirtobrutinib Matched Placebo | Treatment C: 400 mg Moxifloxacin
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/31 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/31 | 0/30
Other Adverse Events (participants affected / at risk) | 6/30 | 1/31 | 1/30
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment A: 900 mg Pirtobrutinib (N=30) | Treatment B: 900 mg Pirtobrutinib Matched Placebo (N=31) | Treatment C: 400 mg Moxifloxacin (N=30)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 5 (5) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2020-12-01): https://cdn.clinicaltrials.gov/large-docs/21/NCT06215521/Prot_000.pdf
  • Statistical Analysis Plan (2021-02-22): https://cdn.clinicaltrials.gov/large-docs/21/NCT06215521/SAP_001.pdf